CLINICAL TRIAL: NCT01884740
Title: Phase I/II Trial Of Super-Selective Intraarterial Infusion Of Erbitux (Cetuximab) And Avastin (Bevacizumab)For Treatment Of Relapsed/Refractory Intracranial Glioma In Patients Under 22 Years Of Age
Brief Title: Intraarterial Infusion Of Erbitux and Bevacizumab For Relapsed/Refractory Intracranial Glioma In Patients Under 22
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was prematurely closed in December 2021 due to low accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1202012214
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Glioblastoma Multiforme; Fibrillary Astrocytoma of Brain; Glioma of Brainstem; Anaplastic Astrocytoma; Pilomyxoid Astrocytoma; Mixed Oligodendroglioma-Astrocytoma; Brain Stem Glioma; Diffuse Intrinsic Pontine Glioma
Keywords: GBM; AA; FA; PXA; AOA; High grade glioma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SIACI of Erbitux and Bevacizumab (Experimental): Superselective Intraarterial Cerebral Infusion (SIACI) of Erbitux (200 mg/m^2) and Bevacizumab (15 mg/kg)
  Interventions: Drug: SIACI of Erbitux and Bevacizumab

INTERVENTIONS:
Drug: SIACI of Erbitux and Bevacizumab — Subjects will receive a single intra-arterial dose of Cetuximab (200 mg/m^2) and Bevacizumab (15 mg/kg) via Superselective Intraarterial Cerebral Infusion (SIACI).
  Other Names: Cetuximab; Avastin

SUMMARY:
Central nervous system (CNS) malignancies are the second most common malignancy and the most common solid tumor of childhood, including adolescence. Annually in the United States, approximately 2,200 children are diagnosed with CNS malignancy and rates appear to be increasing. CNS tumors are the leading cause of death from solid tumors in children. Survival duration after diagnosis in children is highly variable depending in part on age at diagnosis, location of tumor, and extent of resection; however, most children with high grade glioma die within 3 years of diagnosis. All patients with high grade glioma experience a recurrence after first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. It is unknown if currently used intravenous (IV) therapies even cross the blood brain barrier (BBB). We have shown in previous phase I trials that a single Superselective Intra-arterial Cerebral Infusion (SIACI) of Cetuximab and/or Bevacizumab is safe for the treatment of recurrent glioblastoma multiforme (GBM) in adults, and we are currently evaluating the efficacy of this treatment. Therefore, this phase I/II clinical research trial is an extension of that trial in that we seek to test the hypothesis that intra-arterial Cetuximab and Bevacizumab is safe and effective in the treatment of relapsed/refractory glioma in patients <22 years of age. We expect that this project will provide important information regarding the utility of SIACI Cetuximab and Bevacizumab therapy for malignant glioma in patients <22 years of age and may alter the way these drugs are delivered to our patients in the near future.

DETAILED DESCRIPTION:
The experimental aspects of this treatment plan will include:

1. Subjects will first be treated with Mannitol prior to chemotherapy infusion (Mannitol 25%; 10 mL over 2 minutes) in order to disrupt the blood brain barrier. This technique has been used in several thousand patients in previous studies for the IA delivery of chemotherapy for malignant glioma. We have used this without complication in our patients from our Phase I protocols as well.
2. To treat patients <22 years of age with recurring or relapsing glioma with a single intraarterial delivery (SIACI) of Cetuximab and Bevacizumab. Our Phase I trials have demonstrated the safety of SIACI delivery of these drugs in adults. This trial will focus on the safety and efficacy in patients <22 years of age.

ELIGIBILITY:
Inclusion:

1. Male or female patients, under 22 years of age, with a documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), fibrillary astrocytomas (FA), pilomyxoid astrocytoma (PXA), oligodendroglioma, or anaplastic mixed oligoastrocytoma (AOA), or radiologically diagnosed brainstem glioma
2. Patients must have at least one confirmed and evaluable tumor site.

   *A confirmed tumor site is one in which is biopsy-proven with the exception of brainstem glioma which will be eligible with radiographic diagnosis. NOTE: Radiographic procedures (e.g., Gd-enhanced MRI or CT scans) documenting existing lesions must have been performed within three weeks of treatment on this research study.
3. Patients must have a Karnofsky or Lansky performance status 70%. Karnofsky is used for patients older than or equal to the age of 16 years and Lansky for those under 16 years old and an expected survival three months.
4. No chemotherapy for three weeks prior to treatment under this research protocol and no external beam radiation for eight weeks prior to treatment under this research protocol.
5. Patients must have adequate hematologic reserve with absolute neutrophils greater than or equal to 1000/mm3 and platelets greater than or equal 100,000/mm3.
6. Pre-enrollment chemistry parameters must show: bilirubin less than 1.5X the institutional upper limit of normal (IUNL); AST or ALT less than 2.5X IUNL and creatinine less than 1.5X IUNL.
7. Pre-enrollment coagulation parameters (PT and PTT) must be less than 1.5X the IUNL.
8. Concomitant Medications:

   Growth factor(s): Must not have received within 1 week of entry onto this study.

   Steroids: Systemic corticosteroid therapy is permissible in patients with CNS tumors for treatment of increased intracranial pressure or symptomatic tumor edema. Patients with CNS tumors who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to study entry.
9. Patients of reproductive age must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
10. Patients or their parents/guardians must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.
11. Because of known concerns with Avastin and wound healing, craniotomy patients are eligible for the treatment if they have had a craniotomy greater than two weeks prior to IA therapy. Craniotomy or major procedure after SIACI Avastin therapy should wait 4 weeks. Minor surgeries may be performed after two weeks.

Exclusion:

1. Previous treatment with Avastin and Cetuximab
2. Females who are pregnant or lactating.
3. Females of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period. If they do not agree, they will be ineligible for the study.
4. Patients with significant concurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Greenfield, MD PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCrea HJ, Ivanidze J, O'Connor A, Hersh EH, Boockvar JA, Gobin YP, Knopman J, Greenfield JP. Intraarterial delivery of bevacizumab and cetuximab utilizing blood-brain barrier disruption in children with high-grade glioma and diffuse intrinsic pontine glioma: results of a phase I trial. J Neurosurg Pediatr. 2021 Aug 6;28(4):371-379. doi: 10.3171/2021.3.PEDS20738. Print 2021 Oct 1. PMID 34359048
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34359048/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SIACI of Erbitux and Bevacizumab
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SIACI of Erbitux and Bevacizumab
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: Overall Survival (OS) will be measured from the date of the first dose of SIACI Cetuximab/Avastin to the date of death.
Time Frame: 2 Years
Measure: Median (Full Range); unit: days
Arm/Group | SIACI of Erbitux and Bevacizumab
Number analyzed (Participants) | 13
days | 185 [41 to 448]

2. Primary Outcome: Composite Overall Response Rate (CORR)
Description: The overall response proportion along with a 95% confidence interval will be estimated via binomial proportions. The investigator will define "evaluable" patients as patients who met eligibility requirements and have initiated therapy.
Time Frame: 6 Months
Population: The data for this outcome was not collected.
Groups:
- SIACI of Erbitux and Bevacizumab: Superselective Intraarterial Cerebral Infusion (SIACI) of Erbitux (200 m/m^2) and Bevacizumab (15 mg/kg)
  SIACI of Erbitux and Bevacizumab: Subjects will receive a single intra-arterial dose of Cetuximab (200 m/m^2) and Bevacizumab (15 mg/kg) via Superselective Intraarterial Cerebral Infusion (SIACI).
Arm/Group | SIACI of Erbitux and Bevacizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: All treatment emergent adverse events will be assessed and graded according to Common Terminology Criteria for Adverse Events (CTCAE)v. 4.0 terminology for severity, duration, and relationship to research protocol treatment.
Time Frame: 28 days
Measure: Number; unit: adverse events
Arm/Group | SIACI of Erbitux and Bevacizumab
Number analyzed (Participants) | 13
adverse events
  Grade 1 | 4
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS will be assessed by Kaplan-Meier survival analysis, assuming adequate follow-up time. PFS will be measured from the date of the first dose of SIACI Cetuximab/Avastin to the date of progression.
Time Frame: 2 Years
Population: The data for this outcome was not collected.
Arm/Group | SIACI of Erbitux and Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 28 days following treatment procedure with the exception of grade 5 adverse events that were followed for a period of 2 years following treatment.
Description: Patients were closely monitored for toxicity. The primary observation period after IA therapy was 28 days. After the 28 day period, the patient started treatment as recommended by patient's neurooncologist. Toxicities were monitored by history, physical examination, blood tests, and chest x-ray as outlined in the protocol. Within the 28 day period, AEs were assessed on day 0, day 1, and 1 month post-procedure. Participants were followed for grade 5 AEs (death) for 2 years.
Arm/Group | SIACI of Erbitux and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 13/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIACI of Erbitux and Bevacizumab (N=13)
Epistaxis (Surgical and medical procedures) | 2 (2) — One additional participant had a history of nosebleeds and was not included in the analysis.
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated early and participant enrollment was low, resulting in a small sample size (N=13). Having a small sample size may reduce statistical reliability and generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT01884740/Prot_SAP_000.pdf